CLINICAL TRIAL: NCT06461637
Title: Stepped Care Treatment for Common Mental Disorders Among Foreign Domestic Helpers: A Pilot Randomized Controlled Trial
Brief Title: Stepped Care Treatment for Common Mental Disorders Among Foreign Domestic Helpers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY034
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Depression, Anxiety
Keywords: depression; anxiety; stepped-care model; randomized controlled trial; foreign domestic helpers
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped Care Mental Health for Foreign Domestic Helpers (SCMH-FDH) (Experimental): Participants in the SCMH-FDH group will receive a 4-step intervention, i.e., Step 1: Self-Help Intervention and Online Peer-Support, Step 2: Group-Based Intervention, Step 3: Guided Self-Help CBT, and Step 4: Referral to mental health professionals.
  Interventions: Behavioral: Stepped Care Mental Health for Foreign Domestic Helpers (SCMH-FDH)
- Care-As-Usual (CAU) (No Intervention): Participants in CAU group will not receive the stepped care intervention but will have access to care based on their needs and preferences.

INTERVENTIONS:
Behavioral: Stepped Care Mental Health for Foreign Domestic Helpers (SCMH-FDH) — The SCMH-FDH intervention consists of 4 steps. Step 1 involves a self-help intervention (through 12 mental health booklets) delivered in 6 sessions and an online peer support group. Those who did not respond to Step 1 will be referred to Step 2 (group-based resilience workshop). The intervention will be also be delivered in 6 weekly sessions lasting 1-1.5-hours. Those who did not respond to Step 2 will be referred to Step 3 (guided self-help cognitive behavioral therapy, CBT) with guidance from a trained therapist. Self-help materials will be provided. The sessions are spread out over six weeks, with each sessions lasting 30-45 minutes. Those who did not respond to Step 3 will be referred to Step 4 (high intensity interventions provided by mental health professionals). Stepping up is determined by the IAPT-minimum data set. If assessment scores after previous treatment exceeds the defined threshold (PHQ-9 ≥ 10 or GAD-7 ≥ 8), then participants need to step up to the next intervention.
  Arms: Stepped Care Mental Health for Foreign Domestic Helpers (SCMH-FDH)

SUMMARY:
The goal of this pilot randomized controlled trials is to assess the effectiveness of the stepped care approach in treating common mental disorders among foreign domestic helpers in Hong Kong and improve their access to evidence-based psychological treatments.

Participants will be required to complete an online consent form. Then, around 240 eligible participants aged 18-65 years with depression (Patient Health Questionnaire-9 [PHQ-9] ≥ 10) and/or anxiety (Generalized Anxiety Disorder-7 [GAD-7] ≥ 8) will be randomly assigned to the intervention and control group in a ratio of 1:1. Participants assigned in the intervention group will recieved the stepped-care mental health intervention while those assigned to the control group will receive care-as-usual. Assessments of depression, anxiety, and insomnia symptoms, as well as work and social adjustment, quality of life, and treatment credibility and acceptability will be conducted at baseline, week 7 (after Step 1), week 14 (after Step 2), week 21 (after Step 3), and week 33 (12-week follow-up). An assessment of barriers to accessing care will also be collected before treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Foreign domestic helpers aged 18 to 65 years;
2. Able to read, write, and speak in English;
3. Have a PHQ-9 score ≥10 and/or GAD-7 ≥8, indicating caseness or a score that can be classified as a clinical case;
4. Have an internet-enabled device (e.g., laptop computer, smartphone, or tablet);
5. willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Meeting DSM-5 diagnosis of a severe mental illness including psychotic or bipolar disorders as determined by the Mini International Neuropsychiatric Interview (MINI-7);
2. Having a medical condition or neurocognitive disorder that may prevent lifestyle modifications based on the research team's clinical knowledge and experience (e.g., at high risk of fall or dietary change is not suitable as recommended by physicians or dietitians);
3. Current serious suicidal risk as assessed by PHQ-9 Item 9 score >2 (referral information to professional mental health services will be provided);
4. Hospitalization or pregnancy;
5. Current participation in any other clinical trial(s);
6. Current psychological treatment for CMD either psychotherapy or unstable medication in the past 2 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire-9 (PHQ-9) | Baseline, week 7 (After Step 1), week 14 (after Step 2), week 21 (after Step 3), and week 33 (12-week follow-up)
  A 9-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of depressive symptoms. It is rated using a 4-point Likert scale from not at all (0), several days (1), more than half the days (2), and nearly every day (3).
Change in the Generalized Anxiety Disorder-7 (GAD-7) | Baseline, week 7 (After Step 1), week 14 (after Step 2), week 21 (after Step 3), and week 33 (12-week follow-up)
  A 7-item questionnaire assessing the severity of anxiety over the past two weeks. It is rated using a 4-point Likert scale not at all (0), several days (1), more than half the days (2), and nearly every day (3).
Change in the Work and Social Adjustment Scale (WSAS) | Baseline, week 7 (After Step 1), week 14 (after Step 2), week 21 (after Step 3), and week 33 (12-week follow-up)
  A 5-item instrument used for assessing work, social and leisure functioning as well as relationship interaction and home management. It is rated on a 9-point scale from 0 (not at all a problem) to 8 (very severely impaired), with combined score ranging from 0 - 40.

SECONDARY OUTCOMES:
Change in the Insomnia Severity Index (ISI) | Baseline, week 7 (After Step 1), week 14 (after Step 2), week 21 (after Step 3), and week 33 (12-week follow-up)
  A 7-item scale designed to evaluate perceived insomnia severity, distress and functional impairment associated with insomnia. It is rated using a 5-point Likert scale from none (0), mild (1), moderate (2), severe (3), and very severe (4) for questions 1 to 3, and very satisfied (0), satisfied (1), moderately satisfied (2), dissatisfied (3), and very dissatisfied (4) for questions 4 to 7.
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline, week 7 (After Step 1), week 14 (after Step 2), and week 21 (after Step 3)
  A 6-item questionnaire assessing treatment credibility, acceptability/satisfaction, and expectations for success. Two subscales, treatment credibility and outcome expectation, make up the instrument. It is scored on a 9-point Likert scale ranging from not at all (1), somewhat (5) and very much (9).
Change in the Short-Form Six-Dimension (SF-6D) | Baseline, week 7 (After Step 1), week 14 (after Step 2), week 21 (after Step 3), and week 33 (12-week follow-up)
  A 6-item instrument measuring health-related quality of life, including physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in the Treatment Acceptability/Adherence Scale (TAAS) | Baseline, week 7 (After Step 1), week 14 (after Step 2), and week 21 (after Step 3)
  A 10-item questionnaire that is rated by a seven-point Likert scale from 1 (disagree strongly) to 7 (agree strongly). It aims at evaluating treatment acceptability and anticipated treatment adherence of clients in the aspects of credibility, expectancy, and distress.
Assessment of the Barriers to Access to Care Evaluation Scale (BACE) | Baseline
  A 30-item scale used to identify key barriers experienced by people accessing mental health services. It is rated using a 4-point Likert scale from not at all (0), a little (1), quite a lot (2), and a lot (3).

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Yan-Yee Ho, Study Chair — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No